CLINICAL TRIAL: NCT07261228
Title: THE DIFFERENCE IN CARBON FOOTPRINT BETWEEN DIAGNOSTIC UPPER GI ENDOSCOPY IN DYSPEPTIC PATIENTS VERSUS THERAPEUTIC UPPER GI BLEEDING
Status: Recruiting | Type: Observational
Sponsor: King Chulalongkorn Memorial Hospital (Other)
Responsible Party: Principal Investigator, Rapat Pittayanon, Assoc. Prof. Dr., King Chulalongkorn Memorial Hospital
Other Study IDs: RP027
Record Dates: First submitted 2025-11-21; First posted 2025-12-03 (Actual); Last update posted 2025-12-03 (Actual); Status verified 2025-06

CONDITIONS: Carbon Footprint in Upper GI Endoscopy; Dyspepsia; Non-variceal Upper Gastrointestinal Bleeding
Keywords: Carbon footprint; Upper GI endoscopy; EGD; Dyspepsia; Non-variceal upper gastrointestinal bleeding
MeSH Terms: conditions — Dyspepsia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Diagnostic upper GI endoscopy: Dyspepsia patient receiving diagnostic upper GI endoscopy
- Therapeutic upper GI endoscopy: Non-variceal upper GI bleeding patient receiving therapeutic upper GI endoscopy

SUMMARY:
The goal of this observational study is to learn about the carbon footprint produced from diagnostic upper GI endoscopy in patients with dyspepsia and therapeutic upper GI endoscopy in patients with non-variceal upper GI bleeding. The main question it aims to answer is:

• How much carbon footprint is generated from upper GI endoscopy Participants are already receiving diagnostic and therapeutic upper GI endoscopy as part of their regular medical care for dyspepsia and non-variceal upper GI bleeding, respectively. The carbon footprint generated from this treatment process is examined.

DETAILED DESCRIPTION:
Healthcare systems are a significant source of greenhouse gas (GHG) emissions. Gastrointestinal endoscopy accounts for the third largest share of GHG emissions among hospital services, after anesthesiology and intensive care units. Upper GI endoscopy is commonly indicated for diagnostic purposes, such as dyspepsia, or for therapeutic purposes, such as upper GI bleeding. Carbon footprint is defined as the total amount of GHG emissions over the life cycle of a service or product. Prior studies have primarily estimated the overall footprint of endoscopy, often including indirect sources such as patient transportation, rather than direct emissions. To date, no studies have compared the carbon footprint between diagnostic and therapeutic upper GI endoscopy.

This study aims to provide a detailed assessment of the direct carbon footprint generated by endoscopic procedures. We hypothesize that therapeutic endoscopy for upper GI bleeding has higher carbon emissions due to longer procedure time, greater energy consumption, and increased use of disposable equipment compared to diagnostic endoscopy for dyspepsia.

This study is an observational study looking at patients with dyspepsia and peptic ulcer bleeding coming to receive diagnostic and therapeutic upper GI endoscopy, respectively. Patients coming to receive an upper GI endoscopy at King Chulalongkorn Memorial Hospital and Sawanpracharak Hospital, Thailand, who are under the inclusion criteria, are asked to get enrolled in the study and have their data recorded. Without any intervention, they will be treated with the standard treatment and investigation for their conditions.

The timeframe for patient enrollment is two months. The carbon footprint produced was calculated from medical equipment and medication used, energy consumption, and equipment reprocessing. The carbon footprint produced was calculated from when the patient entered the endoscopy center until they left the endoscopy center.

Patients with peptic ulcer bleeding will either get treatment with a bipolar hemostasis probe, a hemostasis clip, or argon plasma coagulation. Epinephrine injection can also be used as an adjunctive treatment.

The success rate and complications after treatment in patients with peptic ulcer bleeding will be recorded by follow-up at 72 hours and 30 days after the procedure.

The data recorded in this study are age, height, weight, underlying diseases, history of alcohol consumption, history of smoking, duration of endoscopic procedure, types and locations of peptic ulcer (if any) according to Forrest classification, and the success rate of bleeding stoppage. These data will be used to calculate the carbon footprint produced from upper GI endoscopy.

Categorical data will be processed using the chi-square test. Continuous data will be calculated using mean and standard deviation, and compared using the unpaired t-test and ANOVA test.

ELIGIBILITY:
Inclusion Criteria:

* Patients with dyspepsia or non-variceal upper GI bleeding
* Age 20-80 years
* Body mass index of 30 or less;
* Receiving one of the following procedure during upper GI endoscopy:

For diagnostic endoscopy: Rapid urease test for H. pylori infection For therapeutic endoscopy: stop bleeding with either Argon plasma coagulation or Bipolar hemostasis probe or Hemostasis clip

Exclusion Criteria:

* Platelet < 50,000
* INR > 2.5
* Pregnancy
* History of allergy to IV sedative medication
* Peptic ulcer grade IIc and III according to Forrest classification
* Patient receiving inhalation anesthesia

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Dyspepsia patients and non-variceal upper GI bleeding receiving upper GI endoscopy at King Chulalongkorn Memorial hospital and Sawanpracharak hospital, Thailand
Sampling Method: Non-Probability Sample
Enrollment: 75 (Estimated)
Dates: Start 2025-06-01 (Actual); Primary Completion 2025-08-31 (Actual); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
To quantify the carbon footprint of diagnostic endoscopy for dyspepsia and therapeutic endoscopy for peptic ulcer bleeding | From enrollment to the time that patients leave the endoscopy room
  The primary outcome is to calculate the carbon footprint produced from diagnostic upper GI endoscopy in dyspepsia patients and therapeutic upper GI endoscopy in peptic ulcer patients, focusing on the carbon footprint produced since the patient enter the endoscopy room until they leave the endoscopy room

SECONDARY OUTCOMES:
To compare carbon emissions between diagnostic and therapeutic upper GI endoscopy | From enrollment to the time that patients leave the endoscopy room
To compare emissions across different hemostatic techniques (clips, argon plasma coagulation, bipolar probe), with or without epinephrine. | From enrollment to the time that patients leave the endoscopy room
To evaluate procedural success rates of bleeding stoppage and adverse events (e.g., perforation, post-procedural sepsis) by different techniques | From enrollment to 30 days after treatment
  To evaluate procedural success rates of bleeding stoppage and adverse events (e.g., perforation, post-procedural sepsis) by different techniques (follow up to 30 days after treatment was given to see rate of recurrent bleeding)

CONTACTS AND LOCATIONS:
Locations (2):
- Thailand (2):
  - King Chulalongkorn Memorial Hospital, Bangkok
  - Sawanpracharak Hospital, Nakhon Sawan

IPD SHARING:
Plan to Share IPD: No